CLINICAL TRIAL: NCT01383265
Title: Randomized Controlled Trial (RCT) to Compare Adenoma Detection Rate of Combined Chromoendoscopy (Indigo Carmine) With Water Infusion in Lieu of Air Insufflation (Water Method) vs. Water Method Alone in Screening Colonoscopy
Brief Title: Combined Chromoendoscopy and Water Method for Screening Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Northern California Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: VANCHCS-GI-006
Record Dates: First submitted 2011-06-24; First posted 2011-06-28 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Colon Polyp
Keywords: screening colonoscopy; adenoma; water method
MeSH Terms: conditions — Colonic Polyps; Adenoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water method and chromoendoscopy (Experimental): Combined water method with chromoendoscopy using 0.008% IC solution for screening colonoscopy
  Interventions: Procedure: Water method and chromoendoscopy
- Water method (Active Comparator): Control method will use plain water with the water method for screening colonoscopy
  Interventions: Procedure: Water method

INTERVENTIONS:
Procedure: Water method and chromoendoscopy — Study method will employ a 0.008% IC solution used with the water method for screening colonoscopy
  Other Names: Water method; Chromoendoscopy; Screening colonoscopy
  Arms: Water method and chromoendoscopy
Procedure: Water method — Control method will use plain water with water method for screening colonoscopy
  Other Names: Screening colonoscopy
  Arms: Water method

SUMMARY:
In a RCT in screening colonoscopy subjects, we will determine if chromoendoscopy using a dilute solution of Indigocarmine (IC) delivered by the water method (study method) will improve adenoma detection rate compared with the water method with plain water alone (control method).

DETAILED DESCRIPTION:
Background: Warm water infusion in lieu of air insufflation (water method) improves overall success of screening colonoscopy and our retrospective data indicate a higher adenoma detection rate. Dye spray methods to improve neoplastic polyp detection such as targeted staining or pancolonic chromoendoscopy have been described.

Aim: In a RCT in screening colonoscopy subjects, we will determine if chromoendoscopy using a dilute solution of Indigocarmine (IC) delivered by the water method (study method) will improve adenoma detection rate compared with the water method with plain water alone (control method).

Methods: After informed consent patients undergoing screening colonoscopy will be randomized to be examined by the study or control method. Study method will employ a 0.008% IC solution. Control method will employ plain water. The water method in both study and control groups will be applied as previously described. The colonoscopy will be performed under sedation. Primary outcome measure: adenoma detection rate; secondary outcome: relevant procedure-related variables.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥50 years old
* Male and female patients
* Scheduled for screening colonoscopy
* Consented and accept randomization to study or control method

Exclusion Criteria:

* Patients who decline to participate
* Unable to give informed consent
* Unable to complete questionnaires due to language or other difficulties

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1177 (Actual)
Dates: Start 2010-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Diagnosis of adenoma | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Leung, MD, Principal Investigator — Sacramento VA Medical Center
Locations (1):
- Sacramento VA Medical Center, Mather, California, United States

REFERENCES:
- [Background] Leung JW, Mann SK, Siao-Salera R, Ransibrahmanakul K, Lim B, Cabrera H, Canete W, Barredo P, Gutierrez R, Leung FW. A randomized, controlled comparison of warm water infusion in lieu of air insufflation versus air insufflation for aiding colonoscopy insertion in sedated patients undergoing colorectal cancer screening and surveillance. Gastrointest Endosc. 2009 Sep;70(3):505-10. doi: 10.1016/j.gie.2008.12.253. Epub 2009 Jun 24. PMID 19555938
- [Background] Leung J, Mann S, Siao-Salera R, Ransibrahmanakul K, Lim B, Canete W, Samson L, Gutierrez R, Leung FW. A randomized, controlled trial to confirm the beneficial effects of the water method on U.S. veterans undergoing colonoscopy with the option of on-demand sedation. Gastrointest Endosc. 2011 Jan;73(1):103-10. doi: 10.1016/j.gie.2010.09.020. PMID 21184876
- [Derived] Leung J, Mann S, Siao-Salera R, Ngo C, McCreery R, Canete W, Leung F. Indigocarmine added to the water exchange method enhances adenoma detection - a RCT. J Interv Gastroenterol. 2012 Jul;2(3):106-111. doi: 10.4161/jig.23728. Epub 2012 Jul 1. PMID 23805387